CLINICAL TRIAL: NCT07249359
Title: Effect of Virtual Reality on Dental Anxiety in Children With Mild Intellectual Disability: A Randomized Controlled Trial
Brief Title: Virtual Reality for Dental Anxiety in Children With Mild Intellectual Disability
Acronym: VR-MID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oasi Research Institute-IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC-2794677
Record Dates: First submitted 2025-11-17; First posted 2025-11-25 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Intellectual Disabilities (F70-F79)
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Distraction (Experimental): immersive VR software delivered through Meta Quest 3® headset during dental procedure
  Interventions: Device: Virtual Reality Distraction - immersive VR software delivered through Meta Quest 3® headset during dental procedure
- Control: Monitor-Based Distraction (Active Comparator): cartoon video displayed in front of dental chair
  Interventions: Device: Control: Monitor-Based Distraction

INTERVENTIONS:
Device: Virtual Reality Distraction - immersive VR software delivered through Meta Quest 3® headset during dental procedure — immersive VR software delivered through Meta Quest 3® headset during dental procedure
  Arms: Virtual Reality Distraction
Device: Control: Monitor-Based Distraction — cartoon video displayed in front of dental chair
  Arms: Control: Monitor-Based Distraction

SUMMARY:
Virtual reality (VR) is a promising non-pharmacological approach to reduce dental anxiety in children with neurodevelopmental disorders. This randomized controlled trial compared a VR-based distraction intervention with conventional monitor-based distraction in children aged 11-15 years with mild intellectual disability and moderate dental anxiety undergoing conservative dental treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 11-15; diagnosis of mild intellectual disability (DSM-5)
* Moderate anxiety (Corah DAS 9-12)
* ≥1 decayed tooth requiring conservative treatment under local anesthesia
* Informed consent from parents/legal guardians

Exclusion Criteria:

* no or slight anxiety
* high or severe anxiety
* visual disorders
* neuromuscular comorbidities interfering with cooperation

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Treatment success | Duration of procedure
  Number of patients with completion of restorative dental procedure under local anesthesia within 50 minutes and positive overall treatment experience (dichotomous: success vs. failure)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ass. Oasi Maria SS, Troina, EN, Italy

IPD SHARING:
Plan to Share IPD: Undecided